CLINICAL TRIAL: NCT03443856
Title: Adjuvant Immunotherapy in Patients With Resected Gastric Cancer Following Preoperative Chemotherapy With High Risk for Recurrence (N+ and/or R1): an Open Label Randomized Controlled Phase-2-study
Brief Title: Postoperative Immunotherapy vs Standard Chemotherapy for Gastric Cancer With High Risk for Recurrence
Acronym: VESTIGE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 1707-GITCG; 2018-000406-36 (EudraCT Number)
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Gastric and Esophagogastric Junction Adenocarcinoma
MeSH Terms: interventions — Nivolumab; Ipilimumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- chemotherapy arm (Other): Completion of the perioperative treatment according to the 2016 ESMO guidelines (change of regimen is not allowed).
  Interventions: Other: chemotherapy
- immunotherapy arm (Experimental): Treatment: Nivolumab 1 mg/kg IV Q3W plus Ipilimumab 3 mg/kg IV Q3W for 4 cycles (3 months) followed by nivolumab 240 mg flat-dose IV Q2W for 9 months.Total treatment time 1 year. No chemotherapy.
  Interventions: Drug: Nivolumab and Ipilimumab

INTERVENTIONS:
Drug: Nivolumab and Ipilimumab — Nivolumab 1 mg/kg IV Q3W plus Ipilimumab 3 mg/kg IV Q3W for 4 cycles (3 months) followed by nivolumab 240 mg flat-dose IV Q2W for 9 months.Total treatment time 1 year
  Arms: immunotherapy arm
Other: chemotherapy — Completion of the perioperative treatment according to the 2016 ESMO guidelines (change of regimen is not allowed).
  Arms: chemotherapy arm

SUMMARY:
The primary objective of the trial is to investigate if nivolumab plus ipilimumab given as adjuvant treatment improve disease free survival (DFS) in patients with stage Ib-IVa gastric and esophagogastric junction adenocarcinoma and high risk of recurrence (defined by ypN1-3 and/or R1 status) following neoadjuvant chemotherapy and resection.

Other study objectives:

* To investigate the safety and effect of adjuvant immunotherapy on long term oncologic outcomes and quality of life of patients in the study
* To correlate nutritional status assessment on outcomes and quality of life of patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric, lower esophageal or GE-junction adenocarcinoma (Siewert I-III)
* Subjects must have completed pre-operative chemotherapy with a fluoropyrimidine-platinum containing regimen and macroscopically complete surgery prior to randomization
* Minimal duration of neoadjuvant chemotherapy should be 6 weeks, maximum 12 weeks.
* Total or distal gastrectomy with D2 lymphadenectomy according to ESMO guidelines should have been completed for gastric and junctional Siewert type III cancers. Ivor Lewis or McKeown oesophagectomy with two field lymphadenectomy should have been performed for junctional Siewert type I cancers. For Siewert type II cancers either total gastrectomy with D2-lymphadenectomy or oesophagectomy with two field lymphadenectomy should have been completed. Open, minimal invasive or hybrid surgical approaches are acceptable as long as the requirements above are fulfilled.
* Regardless of the type of surgery a minimum of 15 lymph nodes should have been resected and examined.
* Recovered from surgery and fit for study treatment as assessed by a multidisciplinary team. Surgery should have been completed 2 to 3 months before randomization.
* ypN1-3 status according to current (8th) version of TNM classification system. In case of an ypN0 status patients must meet the inclusion criterion of R1 resection.
* R0 or R1 resection according to current (8th) version of TNM classification system. In case of R0 resection, patients must meet the inclusion criterion of ypN1-3
* WHO performance status score of 0 or 1
* Age ≥ 18 years
* Adequate organ function assessed within 7 days before randomization:
* White blood cell count (WBC) > 2 x 109/L
* Absolute neutrophil count (ANC) > 1.5 x 109/L
* Platelets ≥ 100 x 109/L
* Hemoglobin ≥ 9 g/dL
* Measured/calculated creatinine clearance ≥ 60 mL/min (according to Cockroft-Gault formula).
* Total bilirubin within normal limits (if the patient has documented Gilbert's disease ≤ 1.5 * ULN or direct bilirubin ≤ ULN)
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5ULN
* Cardiac assessment by 12 Lead ECG and if clinically indicated, cardiac function assessment (using either echocardiography or MUGA scan)
* All toxicities (exception alopecia) attributed to prior anti-cancer therapy must have resolved to grade 1 (NCI CTCAE version 4) or baseline before administration of study drug.
* Women of childbearing potential (WOCBP*) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (HCG)) within 24 hours prior to randomization
* Men who are sexually active with an WOCBP must adhere to contraception (condom) during the study and for a period of 7 months after the last dose of the study treatment in the experimental arm and 6 months in the control arm.
* Patients of childbearing / reproductive potential should use highly effective method of birth control measures during the study treatment period and for at least 5 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* R2 resection status
* M1 stage according to current (8th) version of TNM classification system
* Patients who have undergone complete resection of metastases
* Impaired renal, hepatic, cardiac, pulmonary or endocrine status that compromises the eligibility of the patient for postoperative chemotherapy or immunotherapy
* Clinically significant (that is, active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina pectoris, congestive heart failure (New York Heart Association Classification Class ≥ II), or serious cardiac arrhythmia requiring medication
* Subjects with previous malignancies are excluded unless a complete remission or complete resection was achieved at least 5 years prior to study entry. Adequately treated cervical carcinoma in situ, and localized non-melanoma skin cancer are no exclusion criteria, regardless of timepoint of diagnosis.
* Subjects with active, known, or suspected infectious or autoimmune disease
* Patients who have received antibiotics within the last 14 days before randomization are excluded.
* Subjects with Type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (≥ 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Subjects with > Grade 1 peripheral neuropathy
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Prior or concomitant treatment with radiotherapy/radiochemotherapy
* Any positive test result for HBV or HCV indicating acute or chronic infection
* Known history of HIV or known AIDS and, if required by local practice or positive HIV testing at screening
* Known uncontrollable hypersensitivity to the components of cisplatin/oxaliplatin, fluorouracil (5-FU) or capecitabine, epirubicine or docetaxel
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Ongoing or concomitant use of the antiviral drug sorivudine or its chemically related analogs, such as brivudine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 22 months after last patient in
  Disease free survival is defined as the time interval between randomization and the date of disease recurrence or death from any cause, whichever comes first. Patients alive with no disease recurrence are censored at the date of the last follow-up examination. randomization and the date of disease recurrence or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years after last patient in
  Overall survival is defined as the time interval between the date of randomization and the date of death from any cause. Patients who are still alive when last traced are censored at the date of last follow up.
Loco-regional failure rates | 5 years after last patient in
  Local recurrence is defined as evidence of tumor in the anastomotic area. Regional recurrence is defined as evidence of tumor in the locoregional lymph nodes or other surrounding structures apart from the anastomotic site. Death in absence of loco-regional failure will be considered as a competing risk in the estimation of the cumulative incidence of loco-regional failures. Patients who have not had any such event at the time of data analysis will be censored at the date of the last follow-up examination.
Distant failure rates | 5 years after last patient in
  The diagnosis of distant recurrence requires imaging confirmed by pathology. Once recurrence is confirmed, the date of recurrence is the first date when recurrence was suspected.
  Distant recurrence is defined as recurrence not considered as local or regional.Death in absence of distant failure will be considered as a competing risk in the estimation of the cumulative incidence of distant failures. Patients who have not had any such event at the time of data analysis will be censored at the date of the last follow-up examination
Rate of adverse events according to NCI-CTCAE | 5 years after last patient in
  All adverse events will be recorded; the investigator will assess whether those events are drug related (reasonable possibility, no reasonable possibility) and this assessment will be recorded in the database for all adverse events. AEs will be collected at baseline from randomization.
  Only the worst grade per CTCAE category will be recorded per cycle. All adverse events must be followed until resolution or stabilization. Adverse Events of Special Interest for ipilimumab and nivolumab requiring a close follow-up were identified as a result of signals observed from previous studies involving the protocol treatments. These events require a close follow-up
Quality of life assessed with the EORTC Quality of Life Questionnaire (QLQ-C30) version 3 | questionnaires will be completed at baseline, week 6, 3 months, 6 months, 9 months, 12 months, 15 months
  Quality of life will be assessed with the EORTC Quality of Life Questionnaire (QLQ-C30) version 3. These include five functional scales (physical, role, emotional, social, and cognitive), three symptom (fatigue, nausea and vomiting and pain) and a global health status/QoL scale and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties). The primary HRQoL endpoints that are considered relevant for this study are global health status/QoL and physical functioning.A difference of 10 points on the 100-point QLQ-C30 scale between the two arms will be considered as clinically relevant

CONTACTS AND LOCATIONS:
Overall Officials: Florian Lordick, Study Chair — Universitaetsklinikum Leipzig-Ambulanzen/Sprechstunden, Leipzig, Germany; Maren Knoedler, Study Chair — Universitaetsklinikum Leipzig-Ambulanzen/Sprechstunden, Leipzig, Germany; Elizabeth Smyth, Study Chair — Cambridge University Hospital NHS - Cambridge, UK
Locations (28):
- Czechia (2):
  - Masaryk Memorial Cancer Institute, Brno
  - University Hospital Hradec Kralove, Hradec Králové
- France (3):
  - CHRU de Lille - Hopital Huriez, Lille
  - Hôpital Privé Jean Mermoz, Lyon
  - Gustave Roussy, Villejuif
- Germany (8):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Kliniken Essen-Mitte, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaets Krankenhaus Eppendorf - Universitaetsklinikum Hamburg-Eppendorf KE - University Cancer Center, Hamburg
  - SLK-Kliniken Heilbronn, Heilbronn
  - Universitaetsklinikum Leipzig-Ambulanzen/Sprechstunden, Leipzig
  - Klinikum Rechts der isar Der Technische Universitaet Muenchen - Klinikum Rechts Der Isar, München
  - Universitaetsklinikum Tuebingen-Uni Kliniken Berg, Tübingen
- Israel (2):
  - Rambam Health Care Campus, Oncology Institute, Haifa
  - Rabbin Medical Centre - Tel Aviv, Tel Aviv
- Italy (3):
  - Azienda Ospedaliera a Papa Giovanni XXIII, Bergamo
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
- Oslo University Hospital - Ullevaal Hospital, Oslo, Norway
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- Spain (4):
  - Institut Catalan d'Oncologia - ICO Badalona, Badalona
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Hospitalario A, Pamplona
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (4):
  - Cambridge University Hospital NHS, Cambridge
  - Royal Marsden Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smyth E, Knodler M, Giraut A, Mauer M, Nilsson M, Van Grieken N, Wagner AD, Moehler M, Lordick F. VESTIGE: Adjuvant Immunotherapy in Patients With Resected Esophageal, Gastroesophageal Junction and Gastric Cancer Following Preoperative Chemotherapy With High Risk for Recurrence (N+ and/or R1): An Open Label Randomized Controlled Phase-2-Study. Front Oncol. 2020 Jan 30;9:1320. doi: 10.3389/fonc.2019.01320. eCollection 2019. PMID 32083013